CLINICAL TRIAL: NCT01925365
Title: Hypocholesterolaemic and Prebiotic Effects of a Whole-grain Oat-based Breakfast Cereal in a Cardio-metabolic 'at Risk' Population
Brief Title: Health Benefits of Whole Grain Oats in Population at Risk of Cardio-metabolic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Jordans Cereals (Biggleswade, UK) (Unknown)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UREC 09/12; University of Reading (Other: Reading University)
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Cardiovascular Disease; Hypercholesterolemia
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wholegrain cereal oats (Experimental): Volunteers had to consume wholegrain cereals oats (WGO)(45g/day) for six weeks followed by a four week wash out period.
  Interventions: Dietary Supplement: wholegrain cereals oats (WGO)
- Non wholegrain cereals (Placebo Comparator): Volunteers had to consume non wholegrain cereals (NWG)(45g/day) for six weeks followed by a four week wash out period.
  Interventions: Dietary Supplement: Non wholegrain cereals

INTERVENTIONS:
Dietary Supplement: wholegrain cereals oats (WGO) — Volunteers had to consume wholegrain cereals oats (WGO)(45g/day) for six weeks followed by a four week wash out period
  Arms: Wholegrain cereal oats
Dietary Supplement: Non wholegrain cereals — Volunteers had to consume non wholegrain cereals (NWG)(45g/day) for six weeks followed by a four week wash out period.
  Arms: Non wholegrain cereals

SUMMARY:
Intake of whole grain cereals has been associated with reducing the risk of hyperlipidaemia and heart disease, however the mechanisms by which oats or oat fractions exert this effect is not totally clear. Furthermore, several large epidemiological studies and a number of recent meta-analyses of nutritional interventions have reported a positive association between increased whole grain intake and reduced risk of developing a range of chronic diseases. Recognising the important role of the gut microbiota in metabolism and metabolic disease risk, we examined the impact of whole grain oats on the human gut microbiota and cardio-metabolic risk factors.

The main aims of this human study is to determine the effectiveness of a low GI whole grain oats breakfast cereal compared to a high GI, refined breakfast cereal to beneficially modulate gut microbiota and its metabolic output, plasma lipids, gut satiety hormones and inflammation markers in an at risk of cardio-metabolic disease population

ELIGIBILITY:
Inclusion Criteria:

* Men and Women (age range 23-64 y)
* BMI of 18-30kg/m2
* Fasting glucose concentration >5.5 but <7.5mmol/L
* Total cholesterol >5.2 but <7.8mmol/L

Exclusion Criteria:

* medical history of heart disease, diabetes mellitus, cancer, pancreatitis or renal disease
* use of lipid lowering drugs, systemic corticosteroids or drugs for regulating hemostasis
* exposure to any investigational agent <42 d before the study
* presence of gastrointestinal disorder or use of a drug likely to alter gastrointestinal motility or nutrient absorption
* history of substance misuse or alcoholism
* current pregnancy, planned pregnancy, or given birth in the past 12 months
* antibiotic treatment 6 weeks previous to study start date
* allergy or intolerance to intervention breakfast cereals components
* smoking

Ages: 23 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Changes in faecal bacteria population | Changes in faecal bacteria populations upon consumption of the test and control cereals . Faecal samples were collected and analysed at 0, 42, 56, 112, 140 days

SECONDARY OUTCOMES:
Faecal short chain fatty acids | High-performance liquid chromatography (HPLC) was performed to determine faecal SCFA concentration. Faecal samples were collected and analysed at 0, 42, 56, 112, 140 days
Changes in plasma lipids | Fasted plasma samples were analysed for determination of triacylglycerol (TAG), total cholesterol (TC), HDL-cholesterol, LDL-cholesterol. Blood plasma samples were collected and analysed at 0, 42, 56, 112, 140 days

OTHER OUTCOMES:
Changes in insulin resistance, PYY and GLP-1 | Fasted plasma samples were analysed for determination of insulin resistance, PYY and GLP-1. Blood plasma samples were collected and analysed at 0, 42, 56, 112, 140 days
Changes in inflammatory markers | Fasted plasma samples were analysed for determination of IL-6, TNF-a while saliva samples were analysed for sIgA and faecal samples for calprotectin. Blood plasma samples and saliva and faecal samples were collected and analysed at 0, 42, 56, 112, 140
Changes in dietary intake | 4-day diet diaries were collected analysed, to determine the macro and micronutrient content of the participant's diets during each intervention arm. Diet diaries were collected at were collected and analysed at 42 and 112 days.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Julie A Lovegrove, BSc, PhD, RNutr, Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Result] Connolly ML, Lovegrove JA, Tuohy KM. In vitro evaluation of the microbiota modulation abilities of different sized whole oat grain flakes. Anaerobe. 2010 Oct;16(5):483-8. doi: 10.1016/j.anaerobe.2010.07.001. Epub 2010 Jul 17. PMID 20624475
- [Result] Connolly ML, Tuohy KM, Lovegrove JA. Wholegrain oat-based cereals have prebiotic potential and low glycaemic index. Br J Nutr. 2012 Dec 28;108(12):2198-206. doi: 10.1017/S0007114512000281. Epub 2012 Feb 24. PMID 22360862
- [Derived] Connolly ML, Tzounis X, Tuohy KM, Lovegrove JA. Hypocholesterolemic and Prebiotic Effects of a Whole-Grain Oat-Based Granola Breakfast Cereal in a Cardio-Metabolic "At Risk" Population. Front Microbiol. 2016 Nov 7;7:1675. doi: 10.3389/fmicb.2016.01675. eCollection 2016. PMID 27872611